CLINICAL TRIAL: NCT03279133
Title: A Pilot/Feasibility Study of Ledipasvir/Sofosbuvir as Treatment for Hepatitis C in Hematopoietic Cell Transplantation (HCT) Recipients.
Brief Title: Ledipasvir/Sofosbuvir Treatment for Hepatitis C in HCT Recipients.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to find eligible patients with untreated hepatitis C virus.
Sponsor: Kaiser Permanente (Other)
Collaborators: City of Hope National Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-337-2116
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — ledipasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Intervention Model Description: This is an open-label pilot, safety, feasibility study to treat candidates for HCT infected with hepatitis C prior to the transplantation to reduce the complications associated with hepatitis C in the post-transplant setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LDV/SOF for 12 weeks. (Experimental): Ledipasvir 90mg/Sofosubvir 400mg fixed-dose combination (FDC) tablet for 12 weeks.
  Interventions: Drug: Ledipasvir 90mg/Sofosubvir 400mg

INTERVENTIONS:
Drug: Ledipasvir 90mg/Sofosubvir 400mg — Ledipasvir 90mg/Sofosubvir 400mg (LDV/SOF) FDC is to be administered once daily with or without food for12 weeks.
  Other Names: Harvoni

SUMMARY:
The prevalence of Hepatitis C Virus (HCV) infection was reported to range between 10% and up to 30% prior to institution of routine HCV screening in recipients of HCT (hematopoietic cell transplantation). In an Italian prospective study 6% of HCT candidates were positive for HCV RNA. HCV in recipients of HCT carries both short-term and long-term consequences. In the short-term those with HCV after hematopoietic cell transplantation have been associated with risk for sinusoidal obstruction syndrome especially in patients with some level of hepatic dysfunction going in to the transplant. In addition, the type of conditioning chemotherapy (e.g., busulfan) and radiation may increase risk for sinusoidal obstruction syndrome. The rate of hematopoietic recovery was found to be lower in HCV infected recipients, with delayed neutrophil and platelet engraftment.

In the long-term, HCV may flare up once immunosuppression is being tapered off. The issue of reactivation of viral hepatitis (HBV and HCV) after HCT has been well documented. The risk for HCV reactivation in allogenic HCT in one study was reported at 100% by 12 months after HCT, with risk for death related to HCV of 8%. Also, of concern is rapid progression of liver disease in long-term survivors of HCV+ HCT. In such patients, cumulative incidence of cirrhosis has been reported in up to 11% and 24% at 15 and 20 years after HCT respectively.

Hepatitis C infection is associated with significant morbidity and mortality, due to the short-term and long-term complications associated with it. Treatment of hepatitis C virus with direct-acting antiviral (DAA) agents pre-hematopoietic cell transplantation (HCT) in candidates with hepatitis C may lead to reduction of both short-term and long-term complications from it.

Treatment with DAA's pre-HCT in candidates with hepatitis C would potentially prevent complications of hepatitis C infection; prevent reactivation of hepatitis C post-HCT, prevent delay in hematopoietic recovery (especially neutrophils and platelet), possibly reduce risk for sinsusoidal obstruction syndrome, prevent relapse of malignancy that could be related to hepatitis C (non-Hodgkin lymphoma), reduce non-relapse mortality and long-term complications (cirrhosis).

DETAILED DESCRIPTION:
This is an open-label observational/ feasibility study to treat candidates for HCT infected with hepatitis C prior to the transplantation to reduce the complications associated with hepatitis C in the post-transplant setting.

The study will be conducted at Kaiser Permanente Los Angeles Medical Center and City of Hope National Medical Center, Duarte, CA.

There is no data available on the outcomes of treating hepatitis C with DAA's pre-HCT in candidates with hepatitis C infection. The ASBMT task force made recommendation to consider treating hepatitis C infection pre-HCT based on potential benefits it may be associated with. A single case report has documented benefit of treating a donor infected with hepatitis C prior to stem cell collection with DAA and ribavirin

Subject Population will include autologous or allogeneic HCT candidates (for hematologic malignancy) who have hepatitis C infection. Subjects will be considered treatment-experienced if they have received prior interferon-based therapy. Treatment-experienced patients with prior use of DAA(s) are excluded from study participation.

This study will treat HCV patients prior to HCT, with the goal of reducing early post HCT complications in the first 100 days post HCT followed by measuring outcomes at 2 years post HCT.

Subjects will receive LDV 90mg/SOF 400mg FDC for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be male or female at least 18 years of age at time of screening
2. Participant must be able to provide written Informed Consent
3. Participant must be able to adhere to study visit/procedure schedule and protocol requirements
4. Time available (at least 12 weeks) for treatment of hepatitis C prior to autologous or allogeneic transplantation
5. First autologous or allogeneic HCT and hematologic disease in remission on initiation of antiviral therapy for hepatitis C infection
6. Patients with myelodysplastic syndrome, aplastic anemia or hemoglobinopathies will be eligible to participate regardless of disease status if plan is to proceed to HCT
7. Female participant without childbearing potential must meet at least one of the following:

   * Postmenopausal defined as women >54 years of age with amenorrhea for ≥ 2 years prior to screening
   * Surgically sterile defined as bilateral tubal ligation or bilateral oophorectomy or hysterectomy
   * Has male sexual partner with vasectomy
8. Female participant of childbearing potential must meet at least one of the following:

   * Must be using at least 1 effective contraceptive method at screening and agree to practice 2 effective contraceptive methods1 for study duration, starting Screening through 30 days after stopping study drug
   * Practice total abstinence from sexual intercourse (minimum 1 complete menstrual cycle)
   * Sexually active with female partner only
9. Male participant who is not surgically sterile and is sexually active with female partner of childbearing potential must agree to practice 2 effective contraceptive methods1 for study duration, starting at Screening through 30 days after stopping study drug
10. Participant must have the following indicator- of chronic hepatitis C virus infection prior to study enrollment:

    • Positive for HCV RNA at the time of screening
11. Participant screening laboratory result must indicate HCV genotype 1, 4, 5 or 6-infection if historical result is not available.

Exclusion Criteria:

1. Participant unwilling to provide written informed consent
2. Participant unwilling to adhere to study visit/procedure schedule and protocol requirements
3. Participant is pregnant or is a breastfeeding female
4. Positive test result for hepatitis B surface antigen (HBsAG), hepatitis B core antibody (HBcAb), or confirmed positive anti-HIV antibody test
5. Received study contraindicated medications prior to study drug administration including but not limited to those listed in the Full Prescribing Information Sheet for ledipasvir/sofosbuvir (Harvoni®).
6. Clinically significant abnormalities or co-morbidities, other than HCV infection that in opinion of the investigator makes subject unsuitable for this study or drug regimen
7. Prior or current use of any investigational or commercially available anti-HCV agents other than interferon or ribavirin or receipt of any investigational product within 6 weeks prior to study drug administration
8. Prior treatment of chronic HCV infection with a direct acting antiviral agent(s): telaprevir, boceprevir, sofosbuvir, simeprevir, or other direct acting antiviral
9. History of solid organ transplant
10. Screening laboratory analyses shows any of the following abnormal laboratory results:

    Estimated Glomerular filtration (eGFR) rate < 30 mL/min
11. Evidence of cirrhosis, documented by one of the following:

    Liver biopsy histologic diagnosis: Metavir Score greater than 3 (includes 3 - 4 or ¾) or Ishak score greater than 4 In the absence of liver biopsy: a FibroScan score greater than or equal to 12.5 kPa or Fibrotest score of >0.75 AND an APRI score greater than 1.5
12. History of liver decompensation: ascites noted on a physical exam, imaging or other test; variceal bleeding; hepatic encephalopathy
13. Confirmed presence of hepatocellular carcinoma indicated on computed tomography, magnetic resonance, or other imaging techniques within 3 months prior to screening
14. HCV genotype performed during screening indicates infection with genotype 2 or 3
15. Recent history of drug or alcohol abuse that could, in the opinion of the investigator, affect adherence to the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-04-29 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of LDV/SOF Treatment in Candidates for HCT with hepatitis C infection | 2 year
  To assess the safety and tolerability/feasibility of the two agent combination, ledipasvir and sofosbuvir (LDV/SOF), through evaluation of toxicities, including type frequency, severity, attribution, time course and duration.

SECONDARY OUTCOMES:
Rate of HCV Relapse Post HCT | 2 Years
  To estimate the rate of hepatitis C relapse post HCT - until 2 year after HCT
Effect of Virologic Suppression on Post HCT Complications | 2 Years
  To evaluate the effect of virologic cure on the short term complications after HCT: hematopoietic recovery (neutrophil and platelet count), liver test abnormality, sinusoidal obstruction syndrome, liver disease decompensation in those with advanced fibrosis
Proportion of Patients with Sustained Virologic Response at Time of Transplant | 2 Years
  To estimate the proportion of patients who attained SVR by the time of transplantation (day 0 of HCT), and remain HCV negative at day 30, day 100, day 180, year 1 and year 2 post HCT
Cumulative Incidence of HCV Relapse | 2 Years
  To estimate the cumulative incidence of hepatitis C relapse
Progression of Liver Fibrosis After Transplant | 2 years
  Monitoring for progression of liver fibrosis post-HCT compared to baseline (prior to initiation of DAA treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Sahota, MD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: Undecided